CLINICAL TRIAL: NCT02202876
Title: Redox Imbalance and the Development of Cystic Fibrosis Diabetes
Acronym: Redoxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Arlene Stecenko, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00060962
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2; Cystic Fibrosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cystic Fibrosis | interventions — Glucose Tolerance Test; Fruit and Vegetable Juices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Aim 1: Children with Cystic Fibrosis (Active Comparator): Cystic Fibrosis children aged 1 to 9 years with normal glucose tolerance receiving Oral Glucose Tolerance Test
  Interventions: Other: Oral Glucose Tolerance Test
- Aim 1: Control Children (Active Comparator): Children with out Cystic Fibrosis aged 1 to 9 years controls with normal glucose tolerance receiving Oral Glucose Tolerance Test
  Interventions: Other: Oral Glucose Tolerance Test
- Aim 2a: Teens with Cystic Fibrosis - High Glycemic Meal (Active Comparator): Cystic Fibrosis subjects 12 years of age or older with normal glucose tolerance eating High Glycemic Index Meal
  Interventions: Other: High Glycemic Index Meal
- Aim 2a: Teens with Cystic Fibrosis - Low Glycemic Meal (Active Comparator): Cystic Fibrosis subjects 12 years of age or older with normal glucose tolerance eating Low Glycemic Index Meal
  Interventions: Other: Low Glycemic Index Meal
- Aim 2b: Cystic Fibrosis Consuming Test Soda (Active Comparator): Participants with Cystic Fibrosis 12 years of age or older with normal glucose tolerance or impaired glucose tolerance consuming a test beverage of a test soda. A week later these participants will have an Oral Glucose Tolerance Test.
  Interventions: Other: Oral Glucose Tolerance Test; Other: Test Soda
- Aim 2b: Cystic Fibrosis Consuming Fruit Juice (Active Comparator): Participants with Cystic Fibrosis 12 years of age or older with normal glucose tolerance or impaired glucose tolerance consuming a test beverage of fruit juice. A week later these participants will have an Oral Glucose Tolerance Test.
  Interventions: Other: Oral Glucose Tolerance Test; Other: Fruit juice

INTERVENTIONS:
Other: Oral Glucose Tolerance Test — 1.75 gm/kg to a maximum of 75 gm of an oral glucose solution
  Other Names: OGTT
  Arms: Aim 1: Children with Cystic Fibrosis; Aim 1: Control Children; Aim 2b: Cystic Fibrosis Consuming Fruit Juice; Aim 2b: Cystic Fibrosis Consuming Test Soda
Other: High Glycemic Index Meal — isocaloric breakfasts - set the high glycemic index to 80
  The nutrient composition of each meal will be 10 kcal per kg, 50% kcal from carbohydrates, 20% kcal from protein, and 30% kcal from fat
  Arms: Aim 2a: Teens with Cystic Fibrosis - High Glycemic Meal
Other: Low Glycemic Index Meal — isocaloric breakfasts - set the low glycemic index to 30
  The nutrient composition of each meal will be 10 kcal per kg, 50% kcal from carbohydrates, 20% kcal from protein, and 30% kcal from fat
  Arms: Aim 2a: Teens with Cystic Fibrosis - Low Glycemic Meal
Other: Test Soda — Test soda containing 60% fructose and 40% glucose at a dose of 1.75 grams per kilogram body weight to a maximum of 75 grams.
  Arms: Aim 2b: Cystic Fibrosis Consuming Test Soda
Other: Fruit juice — Fruit juice containing a combination fructose, glucose, and sucrose at a dose of 1.75 grams per kilogram body weight to a maximum of 75 grams
  Arms: Aim 2b: Cystic Fibrosis Consuming Fruit Juice

SUMMARY:
Cystic fibrosis-related diabetes (CFRD) occurs in almost 20% of teens and 50% of adults. The investigators' long term goal is to determine the cause of CFRD in order to translate this knowledge into therapies aimed at preventing CFRD. Since CFRD and type 2 diabetes share several clinical features and since oxidative stress is a key factor in the development of type 2 diabetes, the investigators explored the role of oxidative stress in CFRD. The investigators discovered a unique CF biochemical signature that they believe could be implicated in the development of CFRD. The investigators found that glucose ingestion in CF teens and young adults causes an acute and profound systemic redox imbalance to the oxidizing state. The degree of redox imbalance was quite severe and would be expected to damage the insulin producing cells as these cells are particularly vulnerable to oxidative stress. Thus, these findings could prove to be a critical factor in the pathogenesis of CFRD. This proposal will test the hypothesis that glucose-induced redox imbalance is an intrinsic, metabolic defect in CF. In addition, because CF people are required to consume a high calorie diet to maintain their weight, the investigators also hypothesize that certain high caloric foods will recapitulate the redox imbalance induced by ingesting glucose and thus hasten the development of CFRD. Specifically, the investigators aim to:

* Determine whether young children with CF have glucose-induced redox imbalance
* Determine whether eating a meal with a high glycemic index induces acute redox imbalance
* Determine whether commonly consumed beverages containing simple sugars (i.e., soda or fruit juice) induce acute redox imbalance

DETAILED DESCRIPTION:
Aim 1: Three groups of subjects will be evaluated: 1. 27 CF children with class I-III mutations aged 1 to 9 years with normal glucose tolerance (NGT), 2. 27 age-matched controls with NGT, and 3. 15 CF children with class IV-VI CF transmembrane conductance regulator (CFTR) mutations ages 1 to 9 years. After obtaining informed consent from the parents, subjects will undergo an overnight fast with nothing to eat or drink except water for 10 hours. The children will be asked to withhold all short-acting bronchodilators prior to the start of the study visit and to withhold all long-acting bronchodilators for a minimum of ten hours prior to the start of the study visit. Prior to the study visit, parents will be given a three-day diet journal in which they will record in detail everything each child consumes during the recording period. Details include amount of food or drink and brand names as well as pancreatic enzyme replacement therapy (PERT) dose given with each meal or snack. The recording period will include two week days and one weekend day. The children will have an intravenous (IV) line placed and blood drawn for measurement of plasma glucose, insulin, and cysteine (CyS)/cystine (CySS) redox state. Then the child will be given 1.75 gm/kg to a maximum of 75 gm of an oral glucose solution to drink and will be coached to drink it within 10 minutes. Blood will be drawn 30 minutes after glucose ingestion for repeat measures of glucose, insulin, and redox status. Blood will be drawn 2 hours after glucose ingestion for repeat measures of glucose, insulin, and redox status. Subjects who completed the protocol will be approached to reconsent and repeat the protocol annually to track their level of glucose intolerance and monitor for conversion to CF Diabetes. For children who are able, exhaled breath condensate (EBC) will also be collected prior to the oral glucose tolerance test (OGTT) and immediately following completion of the 2 hour blood draw. EBC will be analyzed for Cys/CySS redox coupling.

Aim 2a: Forty-four CF subjects 12 years of age or older with NGT or impaired glucose will undergo a meal challenge with half randomized to receive a test meal with a high glycemic index and half a meal with a low index. Subjects will fast overnight for 10 hours taking nothing to eat or drink except water. Subjects will be instructed to withhold all short-acting bronchodilators for a minimum of four hours prior to the start of the study visit and withhold all long-acting bronchodilators for a minimum of ten hours prior to the start of the study visit. Following informed consent, participants will first undergo indirect calorimetry for determination of resting metabolic rate and substrate oxidation; this will occur only in participants 16 years old and older. An intravenous line (IV) will then be inserted; and an iPro sensor placed for continuous glucose monitoring (CGM); placement of the CGM will be optional as our experience with this protocol indicates that some CF patients will not volunteer for CGM placement but will for IV placement. If the iPro sensor is inserted; it must be in place for a minimum of 60 minutes prior to the baseline blood draw to allow the iPro sensor device to detect interstitial glucose levels accurately. Blood will be drawn for measurement of glucose, insulin, Cys/CySS redox status, acylcarnitine, total carnitine, proteomics and metabolomics analysis on subjects 16 years older and older. For the subjects 12 years old to 15 years old, blood will be drawn for measurement of glucose, insulin, Cys/CySS redox status, and proteomics. The subject will then be instructed to eat one of two tests meals in ten minutes. Subjects must complete the meal. Meals will be isocaloric breakfasts with one meal having a high glycemic index and one a low. The nutrient composition of each meal will be 10 kcal per kg, 50% kcal from carbohydrates, 20% kcal from protein, and 30% kcal from fat. Blood will be drawn for repeat measures of glucose, insulin, CyS/CySS redox state1, 2, and 3 hours after the test meal on all subjects. Blood will be drawn for proteomics at base line and at 3 hours on all subjects. Additional blood will be drawn at baseline and 2 hrs after the meal for measurement of acylcarnitine, total carnitine,and metabolomics and biomarkers related to fatty acid metabolism on subjects 16 years old and older. Following the 3 hour blood draw, the IV line and iPro sensor, if placed, will be discontinued. A whole-body dual energy X-ray absorptiometry (DEXA) scan will be administered at the completion of the 3 hr blood draw for analysis of body composition; this test will be performed only on those subjects 16 years old and older. Female participants will be required to complete a urine pregnancy test prior to the DEXA scan to confirm a non-pregnant status. If the participant's urine pregnancy test shows a positive pregnancy, the DEXA scan will not be completed. Following the DEXA scan, the subject will be discharged home. Prior to their study visit, participants16 years and older will be given instructions to complete a 3-day food record for estimation of usual dietary intake as part of their standard CF care.

Aim 2b. Forty-four CF subjects 12 years of age or older with NGT or impaired glucose will initially undergo a test beverage challenge, using a test soda that contains 60% fructose and 40% glucose or fruit juice that contains a combination fructose, glucose, and sucrose at a dose of 1.75 grams per kilogram body weight to a maximum of 75 grams. One to four weeks later all subjects will have an OGTT, that is, ingestion of oral glucose solution at a dose of 1.75 grams per kilogram to a maximum of 75 grams. Of the 44 subjects drinking the test beverage, twenty-two will be administered the soda, and twenty-two will be administered fruit juice Subjects will fast overnight for 10 hours taking nothing to eat or drink except water. Subjects will be instructed to withhold all short-acting bronchodilators for a minimum of four hours prior to the start of the study visit and withhold all long-acting bronchodilators for a minimum of ten hours prior to the start of the study visit. After obtaining informed consent participants will have an intravenous line (IV) inserted. Blood will be drawn for measurements of glucose, insulin, and Cys/CySS redox status at baseline or zero minutes. The subject will then be instructed to drink a test beverage, either a test soda or fruit juice, in ten minutes that was prepared by the research bio-nutritionist. Repeat blood samples will be drawn for measures of glucose, insulin, and CyS/CySS redox state ½ hour, 1 hour and 2 hours from the initial consumption of the test beverage drink. During the study visit a beverage intake questionnaire will be administered to assess the patient's overall intake of sweetened beverages. At the completion of the visit the participant will be scheduled for a subsequent visit in one to four weeks for repeat testing using the same guidelines as above, but the test drink to be used is a glucose solution (glucola) used for the standard OGTT. The 75 gram glucola drink will be used for testing; the dose administered will be determined by multiplying the patients weight x 1.75 grams; the dose administered is not to exceed 75 grams. Subjects must consume all of the drink. Blood samples will be drawn at baseline (prior to glucola intake) and then repeat blood samples will be drawn for measures of glucose, insulin, and CyS/CySS redox state ½ hour, 1 hour and 2 hours from the initial consumption of the glucola drink. Insertion of the continuous glucose monitor is optional during the test beverage challenge and the redox OGTT.

ELIGIBILITY:
Aim 1

Inclusion Criteria:

For CF children with class I-III mutations

* CF diagnosed by pilocarpine electrophoresis sweat test and/or CFTR genetic mutation analysis
* CFTR mutation analysis showing two Class I to III mutations
* Aged 1-9 years
* On a clinically stable medical regimen for at least three weeks
* No IV or oral antibiotics for a respiratory exacerbation for at least three weeks
* No hospitalization for at least six weeks

For CF children with class IV-VI mutations

* CF diagnosed by pilocarpine electrophoresis sweat test and/or CFTR genetic mutation analysis
* CFTR mutation analysis showing at least one Class IV-VI mutation
* Aged 1-9 years
* On a clinically stable medical regimen for at least three weeks
* No IV or oral antibiotics for a respiratory exacerbation for at least three weeks
* No hospitalization for at least six weeks
* Not taking pancreatic enzyme replacement therapy

For age-matched controls

* No acute illness for at least six weeks
* Never been hospitalized except at birth following a full term delivery
* Aged 1 to 9 years
* Without any chronic illness requiring prescription medications

Exclusion Criteria:

* Current or past diagnosis of CFRD (for CF children)
* Parents unwilling to have an IV inserted for blood draws

Aim 2a

Inclusion Criteria:

* CF diagnosed by pilocarpine electrophoresis sweat test and/or CFTR genetic mutation analysis
* CFTR mutation analysis showing two Class I to III mutations
* Aged 12 years or older
* On a clinically stable medical regimen for at least three weeks
* No IV or oral antibiotics for a respiratory exacerbation for at least three weeks

Exclusion Criteria:

* Current or past diagnosis of CFRD
* Allergy or intolerance to egg or dairy products

Aim 2b

Inclusion Criteria:

* CF diagnosed by pilocarpine electrophoresis sweat test and/or CFTR genetic mutation analysis
* CFTR mutation analysis showing two Class I to III mutations
* Aged 12 years or older
* On a clinically stable medical regimen for at least three weeks
* No IV or oral antibiotics for a respiratory exacerbation for at least three weeks
* Subjects who have or have not completed the redox meal challenge are allowed to participate

Exclusion Criteria:

* Current or past diagnosis of CFRD
* Allergy or intolerance to any component of the test beverage (i.e., soda, fruit juice) and glucola

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
Acute oxidation | Up to three hours
  cysteine/cysteine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Stecenko, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No